CLINICAL TRIAL: NCT06970925
Title: Pilot Study Evaluating Efficacy and Economic Advantage of Sucrosomial® Iron Post-operative Supplementation vs Standard of Care in Patients After Cardiac Surgery
Brief Title: Pilot Study Evaluating the Advantages of Sucrosomial® Iron Post-operative Supplementation vs Standard of Care After Cardiac Surgery
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-25-119
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Surgery
MeSH Terms: interventions — sucrosomial iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sucrosomial® Iron (Experimental): Patients will receive iron supplementation with Sucrosomial® Iron
  Interventions: Dietary Supplement: Sucrosomial Iron (SI)
- Iron Sucrose injections. (Active Comparator): Patients will receive standard of care Iron Sucrose injections.
  Interventions: Dietary Supplement: Sucrosomial Iron (SI)

INTERVENTIONS:
Dietary Supplement: Sucrosomial Iron (SI) — The Sucrosomial Iron (SI) you may receive is a considered a supplement, so it has not been approved by the U.S. Food & Drug Administration (FDA) for sale. However, it is available for over-the-counter purchase. Sucrosomial Iron (SI) has been developed by PharmaNutra.

SUMMARY:
Primary objective: to evaluate the non-inferiority in terms of improvement of hemoglobin (Hg) levels within 30 days postoperatively between two proposed treatments.

Secondary objective: to evaluate the financial costs associated with Sucrosomial® Iron treatment compared to Iron Sucrose (IV), while demonstrating non-inferiority in the improvement of hemoglobin levels, reduction in transfusion requirements, and reduction of hospital/ICU stay length

ELIGIBILITY:
Inclusion Criteria:

* ICU hospitalized patients who underwent non-emergent cardiac surgery
* Post operative iron deficient or anemic patients (Hb< 12 for both men and women).
* Patients following the same pre-operative protocol
* Age >18 years

Exclusion Criteria:

* Post operative day 1 Hg <9
* Age >90 years
* Patients with cancer or other chronic conditions that impair erythropoiesis (e.g. MDS)
* Stage 3, 4 renal disease
* Intraoperative transfusion of PRBC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in hemoglobin levels | 30 days
  Delta change of hemoglobin levels assessed at T1 in Sucrosomial Iron group to demonstrate non-inferiority compared to the Standard of Care.
Financial Cost | 30 Days
  Financial costs associated with Sucrosomial® Iron treatment compared to Iron Sucrose (IV)

SECONDARY OUTCOMES:
Transfusion requirements | 30 Days
  Reduction in transfusion requirements, measured by the number of transfusions needed during the study period.
Length of Stay | 30 Days
  Length of hospital stay measured from the date of surgery to discharge. Length of ICU stay measured from date of surgery to date of ICU discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Englewood Hospital, Englewood, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No